CLINICAL TRIAL: NCT04889833
Title: Effects of Hypnosis Therapy on Outcomes in Shoulder Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1.0 - 20203698
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Opioid Use
Keywords: hypnosis; shoulder arthroplasty
MeSH Terms: conditions — Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Therapy Group (Experimental): Patients will receive questionnaires to establish their attitudes/beliefs toward hypnosis, baseline pain, anxiety, & shoulder function. 7 days before surgery, they will receive a pre-recorded video (~19 min) of guided hypnosis to be watched at least 1x/day, until surgery. Before & after the video, they will rate pain/anxiety levels. On the day of surgery, they will watch the video again & answer questions about their average anxiety and pain level. After surgery, they will watch the video each day and report on pain/anxiety, medication use, satisfaction, and sleep disturbance until postoperative day 7. Postoperative course will be otherwise completely standard of care, including a clinic visit at 10 days after surgery, where they will be given these same questionnaires. Patients will answer them again on postoperative day 49, constituting a study endpoint. Access to pain medication & study doctor will be the same as any shoulder arthroplasty patient regardless of study participation.
  Interventions: Behavioral: hypnosis therapy
- Usual Care Group (No Intervention): Patients will receive questionnaires to establish their attitudes/beliefs toward hypnosis, baseline pain, anxiety, & shoulder function. 7 days before surgery, they will receive a daily questionnaire about their pain & anxiety over the last 24 hours. On the day of surgery, before they are given any anesthesia, they will answer questions about their average anxiety & pain levels. Starting the next morning on the day following surgery and every day for the subsequent week, they will be given questionnaires about their pain & anxiety levels, medication use, satisfaction, and sleep disturbance due to pain. Their postoperative course will be otherwise completely standard of care, including a first postoperative clinic visit at 10 days after surgery, where the patients will be given these same questionnaires. Finally, patients will answer them one more time on postoperative day 49 and this will constitute a study endpoint. The whole process each day should take approximately 10 minutes.

INTERVENTIONS:
Behavioral: hypnosis therapy — Pre-recorded hypnosis therapy audio recording with accompanying visual of a calm ocean to be played at least once daily for 7 preoperative days, the day of surgery, and for 7 days postoperatively.
  Other Names: hypnotherapy
  Arms: Hypnosis Therapy Group

SUMMARY:
The purpose of this study is to collect information to evaluate the role of the psychogenic component of pain induced by anxiety on postoperative outcomes in major orthopaedic surgery and to determine whether hypnosis therapy provided during the perioperative period will lead to decreased use of opioid therapy. Patients are randomly assigned to one of two treatment groups: (I) usual care, or; (II) hypnotherapy treatment. Patients have an equal chance of being assigned to one of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary shoulder osteoarthritis, massive cuff tear arthropathy, and rotator cuff arthropathy requiring a primary total or reverse shoulder replacement,
* the ability to read, speak, and understand English
* the ability and willingness to use a web-based application (OBERD) on a smartphone, pad, or computer, and
* 18 years of age or older.

Exclusion Criteria:

* shoulder replacement for the treatment of acute proximal humerus fractures
* hemiarthroplasty
* revision shoulder replacement
* patients with active cancer or receiving palliative care
* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Perioperative Anxiety | 7 days before surgery, day of surgery, 7 days after surgery
  Patient-reported anxiety in the perioperative period
Change in Perioperative Pain | 7 days before surgery, day of surgery, 7 days after surgery
  Patient-reported pain in the perioperative period
Change in Opioid Consumption | 7 days after surgery, postoperative day 10, postoperative day 49
  Patient-reported opioid consumption in the perioperative period

SECONDARY OUTCOMES:
Change in Anxiolytic Consumption | 7 days after surgery, postoperative day 10, postoperative day 49
  Patient-reported opioid consumption in the perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frankle, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (1):
- Florida Orthopaedic Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No